CLINICAL TRIAL: NCT03254615
Title: Effectiveness of the Numerous Educational Strategy Interventions Seeking to Increase the Percentage of Water Consumed Among Early Elementary School Students With a 1-year Follow up
Brief Title: Effectiveness of the Numerous Educational Strategy Interventions Seeking to Increase the Water Consume in Child
Acronym: ECCA001LCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jose Francisco Gonzalez-Zamora (Other Government)
Responsible Party: Sponsor-Investigator, Jose Francisco Gonzalez-Zamora, M.D. MSc, National Institute of Pediatrics, Mexico
Organization: National Institute of Pediatrics, Mexico (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 016/2017
Record Dates: First submitted 2017-08-08; First posted 2017-08-18 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Water Consumption; Healthy Lifestyle; Elementary School
Keywords: Plain water; Educative strategies; Effectiveness

STUDY DESIGN:
Intervention Model Description: Experimental, analytical, longitudinal, and prospective designs will be employed. The assignment will be conducted by each school.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group I will receive "I Prefer Plain Water" only during the first grade
  Interventions: Behavioral: "I Prefer Plain Water"
- Group 2 (Experimental): Group II will receive "I Prefer Plain Water" during first and second grades
  Interventions: Behavioral: "I Prefer Plain Water"
- Group 3 (Experimental): Group III will receive "I Prefer Plain Water" during first, second, and third grades
  Interventions: Behavioral: "I Prefer Plain Water"

INTERVENTIONS:
Behavioral: "I Prefer Plain Water" — The students will receive four educational sessions of approximately 1 hour. These sessions will be given every 2 weeks, and some will be supervised by a nutritionist.

SUMMARY:
The current project seeks to evaluate the effectiveness of numerous educational strategy interventions to increase the percentage of water consumed among early elementary school students over a 1-year period.

DETAILED DESCRIPTION:
A community intervention trial will be conducted at four public elementary schools of the Coyoacan Delegation in Mexico City. It will include healthy first graders during the 2017-2018 school year whose parents agree to participate through verbal informed consent and a signed privacy notice. These parents will complete a baseline 3-day beverage record (two weekdays and one weekend day). The four schools will be assigned to one of three groups: Group I will receive the educational strategy during the first grade; Group II will receive it during first and second grades; and Group III will receive it during the first, second, and third grades. All schools will have water dispensers inside the classrooms, and the children will receive a reusable 600-mL bottle so they are able to consume water on demand throughout the day. A second record of beverage consumption will be obtained by completing multiple interventions within each group, and a third record will be completed 1 year later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Both girls and boys
* Children whose parents agree to participation in the study through verbal informed consent
* Children whose parents sign a privacy notice

Exclusion Criteria:

* Children who present with any pathology that interferes with the free consumption of water or with the proper execution of the study
* Children for whom it is not possible to obtain a baseline record of beverage consumption

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 329 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of water consumed | Up to 4 years, baseline measurement and once a year
  Changes in average water consumption/ total liquid consumption
Water consumption | Up to 4 years, baseline measurement and once a year
  Changes in the average of water consumption per child over a 3-day period
Total liquid Consumption | Up to 4 years, baseline measurement and once a year
  Changes in the average of total liquids consumed per child over a 3-day period

SECONDARY OUTCOMES:
Effectiveness of educational strategy | Up to 4 years, baseline measurement and once a year
  Changes in the percentage of water consumed, 1 year after completing the interventions within each group relative to baseline measurement

OTHER OUTCOMES:
BMI | Up to 4 years, baseline measurement and once a year
  Indicator of the relationship between weight and height
Health condition | Up to 4 years, baseline measurement and once a year
  Health condition that (in the opinion of the investigator) enables the participant to have free consumption of water
Water consumption per school | Up to 4 years, baseline measurement and on monthly bases
  Quantity of water consumed in 1 month per participating school

CONTACTS AND LOCATIONS:
Overall Officials: Jose F Gonzalez-Zamora, MD MSc, Principal Investigator — Instituto Nacional de Pediatria
Locations (1):
- Instituto Nacional de Pediatria, Mexico City, Coyoacan, Mexico

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/15/NCT03254615/Prot_SAP_000.pdf